CLINICAL TRIAL: NCT05990413
Title: Comparison of Activity Levels of Periscapular Muscles During Open and Closed Kinetic Chain Activities in Individuals With Stroke
Brief Title: Periscapular Muscle Activation During Open and Closed Kinetic Chain in Stroke
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Çiçek Günday, Principle Investigator, Istanbul University - Cerrahpasa
Other Study IDs: 26032023
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Hemiplegia
Keywords: Hemiplegia; Scapular muscles; Muscle timing; Muscle activation; Kinetic chain
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hemiplegic Participants: Participants will be evaluated in terms of inclusion criteria, and fugl-meyer upper extremity performance assessment will be applied to eligible patients and it will be clarified whether they can be included. Participants who may be included in the study will fill in the patient demographic information form prepared by the researchers as a face-to-face interview. This form will take approximately 5 minutes, during which time the muscles will be rested. Then, the viscoelastic properties of the determined muscles of the participants will be evaluated. Finally, the participants will be evaluated in terms of the activation timing and percentages of the muscles determined during an open and closed kinetic chain activity. Half of the participants will do the open kinetic chain activity before the closed kinetic chain activity with a five-minute resting period between activities. The others will start with the closed kinetic chain activity first and then the open kinetic chain activity.
- Healthy Participants: Participants will be evaluated in terms of inclusion criteria. Eligable participants will fill in the patient demographic information form prepared by the researchers as a face-to-face interview. This form will take approximately 5 minutes, during which time the muscles will be rested. Then, the viscoelastic properties of the determined muscles of the participants will be evaluated. Finally, the participants will be evaluated in terms of the activation timing and percentages of the muscles determined during an open and closed kinetic chain activity. Half of the participants will do the open kinetic chain activity before the closed kinetic chain activity with a five-minute resting period between activities. The others will start with the closed kinetic chain activity first and then the open kinetic chain activity.

SUMMARY:
The goal of this observational study is to compare the activity levels of the periscapular (levator scapula, serratus anterior, infraspinatus, upper, middle and lower trapezius) muscles during open and closed kinetic chain activities in individuals with stroke. It is also aimed to reveal the relationship between the timing and percentage of scapular muscle activation, the viscoelastic properties of these muscles, motor performance and capacity. The main questions it aims to answer are:

* The activation timing, percentage and viscoelastic properties of the periscapular muscles of stroke individuals compared to healthy individuals;
* The activation timing and percentages of periscapular muscles during closed kinetic chain and open kinetic chain activities in stroke individuals;
* The relationship between muscle activation timing, muscle activation percentage, viscoelastic properties, upper extremity motor performance and capacity.

The study will include both hemiplegic (n=10) and healthy (n=10) participants. All of the participants will be assessed in terms of scapular muscle activation timing and percentage (with superficial electromyography) during both open kinetic chain and closed kinetic chain activities.

viscoelastic properties of muscles (Miyoton) will be evaluated. Upper extremity movement frequency and quality (MAG-28) and functional performance (Fugl-Meyer) will be evaluated to reveal the status of stroke individuals.

In the study, it is also aimed to reveal the relationship between the timing and percentage of scapular muscle activation, the viscoelastic properties of these muscles, motor performance and capacity. 10 healthy and 10 hemiplegic individuals are planned to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

Stroke patients will be considered eligible for participation if they:

* were at least 6 weeks after stroke (hemorrhagic or ischemic);
* had mild to moderate upper limb motor impairment (score of ≥30 on the Fugl-Meyer upper limb motor part;
* had a negative Neer impingement test;
* could sit or stand up independently at least 10 minutes.

Healthy controls will be considered eligible for participation if they:

* had no self-reported shoulder pain;
* had a negative Neer impingement test.

Exclusion Criteria:

Participants will be excluded according to these criteria:

* being involuntary to participate and unable to follow the instructions;
* being younger than 18 years old;
* body mass index equal or higher than 30;
* shoulder and/or neck pain in the last six months;
* known history of shoulder dislocation, fracture or surgery;
* other systemic and/or neurologic diseases. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The total number of participants participating in the study is planned to be twenty. It is planned that ten of those twenty participants will be healthy as the controls and ten of them will be individuals with hemiplegia as cases.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Muscle activation timing and percentage | 1 day
  Noraxon Surface Electromyography System will be used to assess muscle activation timing and percentage of upper, middle and lower trapezius, serratus anterior, infraspinatus, levator scapulae of all participants. The placement of electrodes will be done according to SENIAM's European Recommendations for Surface Electromyography. Synchronized video capture will be used to determine the phases of the scapular motion during the open and closed kinetic chain exercises (OKC and CKC, respectively). To take the measurement during OKC, participants will be seated in a chair that will support the waist and back, with the feet in contact with the ground. They will be asked to cross the fingers of both hands and to raise both arms overhead as high as they can. For CKC, they will be asked to stand next to a table at level of SIAS and place their forearms on table with the elbows flexed. They will be asked to extend the elbow of the non-measuring arm while shifting body weight to the other side.
Viscoelastic properties | 1 day
  Myoton®PRO Digital Palpation Device will be used to measure the muscle tone, stiffness, and elasticity of muscles below. The patient will be seated with the flexed elbow supported by a pillow next to the body. Measurements will be repeated 3 times.
  * Upper Trapezius: the end-points of a line connecting the spinous process of C7 and the acromion, distally, from the mid-point of the muscle belly
  * Middle Trapezius: the mid-point of a line connecting T4 spinous process to the medial border of spina scapula
  * Lower Trapezius: The mid-point of a line connecting the spinous process of T6 to the medial border of spina scapula
  * Serratus anterior: a- Over the fourth rib, at the midpoint between the latissimus dorsi and the pectoralis major; b- Over the seventh rib, in the midline of the axilla
  * Infraspinatus: Two fingers breadth below the center spine of the scapula
  * Levator Scapulae: Between the posterior margin of SCM and anterior margin of the UT, at level of C4/5

SECONDARY OUTCOMES:
Upper extremity motor performance | 1 day
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. It will be used for the participants only with hemiplegia.

CONTACTS AND LOCATIONS:
Overall Officials: Kubra Kardeş, PT,MSc,PhD-c, Study Chair — Istinye University; Çiçek Günday, PT,MSc,PhD-c, Principal Investigator — Istanbul University - Cerrahpasa; Ayse Zengin Alpözgen, PT,MSc,PhD, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istinye University Physiotherapy and Rehabilitation Reasearch and Application Center, Istanbul, Turkey (Türkiye)